CLINICAL TRIAL: NCT02139631
Title: Evaluation of the Hemodynamic Repercussions of Non Invasive Ventilation in Healthy Individuals by Doppler Echocardiography
Brief Title: Hemodynamic Repercussions of Noninvasive Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Uberlandia (Other)
Responsible Party: Principal Investigator, Gabrielle Silva Vinhal, Avaliação das repercussões hemodinâmicas com o uso de ventilação mecânica não invasiva em indivíduos saudáveis por meio do ecodopplercardiograma, Federal University of Uberlandia
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: 070490
Record Dates: First submitted 2014-04-30; First posted 2014-05-15 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2015-09

CONDITIONS: Haemodynamic Rebound
Keywords: hemodynamic; mechanical ventilation; respiration with positive pressure
MeSH Terms: interventions — Noninvasive Ventilation; Continuous Positive Airway Pressure; Positive-Pressure Respiration

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Healthy volunteers (Experimental): The volunteers initially underwent a clinical examination, spirometry and echocardiography to prove the health state. Then, different levels of positive end expiratory pressure (PEEP) is applied by the noninvasive ventilation in all individuals and the hemodynamic repercussions are evaluated by the doppler echocardiography
  Interventions: Other: Noninvasive ventilation

INTERVENTIONS:
Other: Noninvasive ventilation — Assess the hemodynamic repercussions of the positive end expiratory pressure applied noninvasively
  Other Names: Continuos positive airway pressure; Bilevel; Positive end expiratory pressure

SUMMARY:
The noninvasive ventilation (NIV) is a method of ventilatory support that does not require artificial airway. Its application is associated with complex hemodynamic repercussions, therefore is important to identify them for safety and effectiveness of the technique application.

The main objective of this research is to evaluate the hemodynamic repercussions using doppler echocardiography in healthy volunteers submitted a different values of positive end expiratory pressure (PEEP) by the following ventilatory modes: Continuous positive airway pressure (CPAP) and Bilevel.

The study hypothesis is that the positive end expiratory pressure (PEEP) may cause hemodynamic repercussions as: reduction of the ventricles pre-load, left ventricle after load, cardiac output and reduction in the diameter of the superior vena cava, due to the increase in the intrathoracic pressure and pulmonary volumes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals
* Age between 18 and 40 years old
* Non smoker

Exclusion Criteria:

* Clinical signs or symptoms of any disease decompensation
* History of blood pressure variations by autonomic dysfunction
* Sense of claustrophobia
* Smoker

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-05; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Hemodynamic repercussions of different levels of positive end expiratory pressure applied noninvasively, measured by echocardiography | 5 minutes
  The hemodynamic variables evaluated are: ventricular preload, left ventricle afterload, cardiac output, blood pressure and the vena cava's diameter. All variables will be assessed by echocardiography

SECONDARY OUTCOMES:
Measurement of cardiac output as a predictor of cardiopulmonary adaptation to different pressures. | 5 minutes

OTHER OUTCOMES:
Difference between the hemodynamic effects generated by ventilation modes CPAP and Bilevel | 3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Celia R Lopes, Principal Investigator — Federal University of Uberlandia
Locations (1):
- Federal University of Uberlandia, Uberlândia, Minas Gerais, Brazil

REFERENCES:
- [Result] Pinsky MR. Heart lung interactions during mechanical ventilation. Curr Opin Crit Care. 2012 Jun;18(3):256-60. doi: 10.1097/MCC.0b013e3283532b73. PMID 22473256
- [Result] Grace MP, Greenbaum DM. Cardiac performance in response to PEEP in patients with cardiac dysfunction. Crit Care Med. 1982 Jun;10(6):358-60. doi: 10.1097/00003246-198206000-00002. PMID 7042203
- [Result] Jardin F, Farcot JC, Boisante L, Curien N, Margairaz A, Bourdarias JP. Influence of positive end-expiratory pressure on left ventricular performance. N Engl J Med. 1981 Feb 12;304(7):387-92. doi: 10.1056/NEJM198102123040703. PMID 7005679
- [Result] Schmidt GA. Cardiopulmonary interactions in acute lung injury. Curr Opin Crit Care. 2013 Feb;19(1):51-6. doi: 10.1097/MCC.0b013e32835c35ac. PMID 23201585
- [Result] Fellahi JL, Valtier B, Beauchet A, Bourdarias JP, Jardin F. Does positive end-expiratory pressure ventilation improve left ventricular function? A comparative study by transesophageal echocardiography in cardiac and noncardiac patients. Chest. 1998 Aug;114(2):556-62. doi: 10.1378/chest.114.2.556. PMID 9726745
- [Result] Steingrub JS, Tidswell M, Higgins TL. Hemodynamic consequences of heart-lung interactions. J Intensive Care Med. 2003 Mar-Apr;18(2):92-9. doi: 10.1177/0885066602250369. PMID 15189655